CLINICAL TRIAL: NCT06562777
Title: INvestigating Sex and Gender-Related Differences in Immunotherapy Treatment Effects (INSITE)
Brief Title: Observational Study of Sex Differences in Symptoms During Immune Checkpoint Inhibitor Treatment for People With Cancer
Status: Recruiting | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Deanne Tibbitts, Principal Investigator, OHSU Knight Cancer Institute
Other Study IDs: STUDY00025328; NCI-2023-06611 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00025328 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-08-15; First posted 2024-08-20 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients complete surveys and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-Interventional Study

SUMMARY:
This study aims to learn more about symptoms that patients experience while receiving immunotherapy for cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Characterize sex differences in patient-reported symptomatic immune-related adverse events.

II. Determine the level of discordance between clinician-assessed and patient-reported symptomatic immune-related adverse events according to patient gender.

OUTLINE: This is an observational study.

Patients complete surveys and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older on date of enrollment (Confirmed by review of the date of birth as documented in the Electronic Medical Record (EMR) and subsequently recorded in a CRF.)
2. Histologically confirmed diagnosis of cancer and plan to begin SOC immunotherapy for the treatment of cancer per FDA approval and/or National Comprehensive Cancer Network (NCCN) guidelines (Confirmed by review of cancer diagnosis and treatment plan as documented in the Electronic Medical Record (EMR) and subsequently recorded in a CRF.)
3. Treating oncologist anticipates at least 6 consecutive months of SOC immunotherapy (Confirmed by review of the treatment plan as documented in the Electronic Medical Record (EMR) and subsequently recorded in a CRF.)

Exclusion Criteria:

1. Diagnosed with breast, prostate, testicular, penile, or gynecologic cancer (Confirmed by review of the cancer diagnosis as documented in the Electronic Medical Record (EMR) and subsequently recorded in a CRF.)
2. Previously received immunotherapy (Confirmed by review of cancer treatment history as documented in the Electronic Medical Record (EMR) and subsequently recorded in a CRF.)
3. Life expectancy of <6 months at time of enrollment per the treating oncologist (Confirmed by the professional opinion of the treating oncologist and subsequently recorded in a CRF.)
4. Concurrently receiving a non-immunotherapy treatment, including chemotherapy, biological, or targeted therapy (Confirmed by review of the treatment plan as documented in the Electronic Medical Record (EMR) and subsequently recorded in a CRF.)
5. Concurrently receiving radiation, unless hypofractionated palliative radiation prescribed to alleviate poorly controlled symptoms (e.g. pain) (Confirmed by review of the treatment plan as documented in the Electronic Medical Record (EMR) and subsequently recorded in a CRF.)
6. Participation in a clinical trial of experimental immunotherapy (Confirmed by review of the treatment plan as documented in the Electronic Medical Record (EMR) and subsequently recorded in a CRF.)
7. Needs to rely on a proxy to complete patient-reported outcome instruments (Confirmed by self-report on Health History Questionnaire.)
8. Unwilling or unable to complete consent form and surveys electronically (Confirmed by successful completion of electronic consent form and baseline survey in REDCap.)

Assessment of participant eligibility is at the discretion of the Principal Investigator, Dr. Deanne Tibbitts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will begin standard-of-care (SOC) immunotherapy for the treatment of cancer at OHSU and Knight Cancer Institute Community Hematology Oncology (CHO) clinics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported symptoms | Baseline, weekly thereafter up to 26 weeks
  Will compare the number, severity, and burden of symptoms by sex. Will be assessed using the Common Toxicity Criteria and Adverse Events v1.0 (PRO-CTCAE) reporting tool.
Patient-reported QOL - Part 1 | Baseline, month 3, month 6
  Will use the Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29)
Patient-reported QOL - Part 2 | Baseline, month 3, month 6
  PROMIS Cognitive Function instruments
Patient-reported QOL - Part 3 | Baseline, month 3, month 6
  Selected questions from the EORTC-QLQ-C30 to evaluate the impact of immunotherapy on QOL.
Clinician-assessed patient symptoms | Baseline, month 3, month 6
  Clinicians will rate patient symptoms according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 scoring system, which grades adverse events according to 5 categories of severity and requires evaluation of the extent to which the adverse event can be attributed to treatment ("unrelated" to "definite"). Will examine agreement using intraclass correlations by patient gender.

CONTACTS AND LOCATIONS:
Overall Officials: Deanne Tibbitts, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided